CLINICAL TRIAL: NCT02822638
Title: CoHort of STEMI Patients
Acronym: STEMI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0412
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; biomarkers; STEMI
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In STEMI patient refered for PCI at Louis Pradel Hospital, blood samples were taken on admission at (H0) and 4h after reperfusion.
  To constitute the serum bank of our STEMI cohort, samples were collected the same time as the blood tests done routinely.
  These additional samples were be centrifuged and treated and stored in a collection of biological samples of total serum and plasma and blood at the Biological Resource Center of HCL Neurobiotec at -80 ° C (DC- 2008-72, AC-2013-1867 certified NFS96900 FR13-018140).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI PATIENT Cohort: STEMI PATIENT Cohort
  Interventions: Other: STEMI PATIENT Cohort

INTERVENTIONS:
Other: STEMI PATIENT Cohort — PCI

SUMMARY:
Ischemic heart disease is the leading cause of mortality in industrialized countries. ST elevated acute myocardial infarction is one of its most frequent and deadly manifestation. In the last 20 years, STEMI mortality has been reduced by 50% with the advent of timely reperfusion (primary percutaneous intervention) and significant progression in pharmacologic intervention.

However, death and heart failure incidence after STEMI remain elevated: up to 20% at one year.

Also, therapeutic management following international guidelines is standardized toward a "one-size fits all" therapeutic management.

In order to continue improving myocardial infarction outcomes, there is a need to better understand and individualize therapeutic targets such myocardial reperfusion injury, post reperfusion inflammation, adverse left ventricular (LV) remodeling ….

This knowledge will allow us to propose new therapeutic strategies and in the long run strive towards personalized medicine.

The aim objective of this cohort of STEMI patients is to identify new biological markers of injury and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Diagnosis of STEMI defined by ST segment elevation ≥ 0.2 mV in 2 contiguous leads on a 12-lead ECG.
* Primary PCI within 12 hours of symptoms onset.

Exclusion Criteria:

* Diagnosis of STEMI not confirmed by angiography
* Refusal to participate in the study or to sign the consent
* Inability to give information to the subject about the study
* Lack of medical social coverage
* Deprivation of civil rights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI PATIENT
Sampling Method: Non-Probability Sample
Enrollment: 1204 (Actual)
Dates: Start 2009-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Troponin | Day 0
  Dosage of Troponin at hospital admission and 4 hours after Percutaneous coronary intervention (PCI)
Change in Creatine Kinase | Day 0
  Dosage of Creatine Kinase at hospital admission and 4 hours after PCI

SECONDARY OUTCOMES:
New York Heart Association (NYHA) Class | at admission (Day 0)
Left ventricular ejection fraction (LVEF) | 24 hours after PCI (Day 1)
  LVEF measured by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Michel OVIZE, Pr, Principal Investigator — Centre d'investigation Clinique , Hôpital Cardiovasculaire Louis Pradel 28, Avenue du Doyen Lépine - 69677 BRON
Locations (1):
- Hôpital Cardiovasculaire Louis Pradel 28, Avenue du Doyen Lépine, Bron, France